CLINICAL TRIAL: NCT02041624
Title: An International Non-Interventional Registry on the Quality of Life of Patients With Grass-pollen-induced Allergic Rhinitis Treated With Oralair®.
Brief Title: International Registry on the Quality of Life of Patients With Grass-pollen-induced Allergic Rhinitis
Acronym: ALTO
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Stallergenes Greer (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Other Study IDs: ORA-PES-05-WO
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Allergic Rhinitis Due to Grass Pollens
Keywords: allergic; rhinitis; conjunctivitis; grass pollen; Allergen ImmunoTherapy (AIT); grass mix
MeSH Terms: conditions — Rhinitis; Conjunctivitis

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- allergic rhino-conjunctivitis: Patient with proven allergic rhino-conjunctivitis due to grass pollen

SUMMARY:
The purpose of the present study is to describe patient's perception of quality of life and effectiveness of ORALAIR® over a follow-up period up to 5 years, in real-life settings.

DETAILED DESCRIPTION:
Primary objective:

To describe the patient's perception of the impact of ORALAIR® on his/her health related generic and disease specific quality of life during the grass pollen season in real-life settings.

Secondary objectives:

- To describe the patient's perceived effectiveness of ORALAIR® in allergic rhinoconjunctivitis management in terms of disease intensity, satisfaction and rescue medication

ELIGIBILITY:
Inclusion Criteria:

* Patient of 5 years of age and older at the date of the screening visit
* Patient with proven allergic rhino-conjunctivitis due to grass pollen
* Patient eligible for a grass-pollen Allergen ImmunoTherapy (AIT)
* Patient whose physician prescribed ORALAIR® independently of the study, before the beginning of the grass-pollen season

Exclusion Criteria:

* Patient participating in a clinical trial or in an epidemiological study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with allergic rhino-conjunctivitis are visiting their allergist during grass-pollen season when symptoms are strong. In accordance with the terms of the Marketing Authorization, ORALAIR® treatment has to be set-up "at the right moment" about 4 months before the next grass-pollen season.
Sampling Method: Non-Probability Sample
Enrollment: 740 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | patients will be followed for the duration of the treatment, an expected average of 6 months/year
  The primary objective is to describe the patient's perception of the impact of ORALAIR® on his/her health related generic and disease specific quality of life during the grass-pollen season in real-life settings.

SECONDARY OUTCOMES:
Treatment Effectiveness | patients will be followed for the duration of the treatment, an expected average of 6 months/year
  To describe the patient's perceived effectiveness of ORALAIR® in allergic rhino-conjunctivitis management in terms of disease intensity, satisfaction and rescue medication

CONTACTS AND LOCATIONS:
Overall Officials: Alain DIDIER, MD, Principal Investigator — Hôpital Larrey, Toulouse, France
Locations (1):
- Laboratoire Stallergenes, Antony, France